CLINICAL TRIAL: NCT03093441
Title: A Comparison of High-intensity Interval Training Protocols on Cardiometabolic Markers, Physical Performance, and Psychosocial Markers in College Females
Brief Title: A Comparison of High-intensity Interval Training Protocols on Health and Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Responsible Party: Principal Investigator, Elise Brown, Assistant Professor, Oakland University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OU1002886
Record Dates: First submitted 2017-03-17; First posted 2017-03-28 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: High-intensity interval training; cardiometabolic; physical performance; psychosocial adaptation

STUDY DESIGN:
Intervention Model Description: A parallel-group randomized controlled trial with 9-month follow-up will be conducted. Once initial screening is completed, participants will be randomized into one of three arms: 1) MM-HIIT, 2) R-HIIT, and 3) control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multimodal (Experimental): Multimodal High-Intensity Interval Training Intervention. This group will train using multimodal exercises for 5 sets of 60 seconds of all out work, followed by 3 minutes of rest. Each session will have the same exercises within each set, but every session will be different than the others for movements utilized. There will be three movements used in each set. The first movement will be a strength movement for 4-6 repetitions. The second movement follows the first immediately and is a faster body weight or light implement power movement for 6-8 repetitions. The third movement follows the second immediately and is a very fast, sprint-like movement for the remainder of the 60 seconds. The intent of each set is to be completed with as much effort as possible across the full 60 seconds.
  Interventions: Other: Multimodal High-Intensity Interval Training Intervention
- Rowing (Active Comparator): Multimodal High-Intensity Interval Training Intervention. This group will train using a rowing ergometer for 5 sets of 60 seconds of all out work, followed by 3 minutes of rest (a total of 20 minutes each session). Each training session will be the same across the 12 weeks. The intent of each set is to be completed with as much effort as possible across the full 60 seconds.
  Interventions: Other: Multimodal High-Intensity Interval Training Intervention
- Control (No Intervention): Multimodal High-Intensity Interval Training Intervention. This group will be instructed to continue with any activity they were involved in prior to the study and to not begin any new exercise programs during the course of the study. To incentive participation in this group, the control group will be offered the MM-HIIT intervention the following semester at no cost.

INTERVENTIONS:
Other: Multimodal High-Intensity Interval Training Intervention — The intervention will occur 3 times per week for 12 weeks and include a warm-up, MM-HIIT or R-HIIT training protocol, and a cool down.
  Arms: Multimodal; Rowing

SUMMARY:
Recently, it has been demonstrated that multimodal high-intensity interval training (MM-HIIT) (utilizing resistance-based and functional movements) can produce similar aerobic adaptations compared to high-intensity interval training (HIIT) using rowing but with greater muscle performance in females. In addition, HIIT has been shown to be more enjoyable than continuous training, and this may lead to enhanced self-efficacy and increased physical activity. To the investigators' knowledge, however, the cardiometabolic effects (blood pressure, abdominal/visceral fat, blood sugar, blood lipids/fats) of MM-HIIT have not been reported. The investigators aim to compare MM-HIIT with HIIT using a traditional aerobic fitness exercise (rowing) for the degree of cardiometabolic, physical performance (strength, endurance, power), and psychosocial (self-efficacy and enjoyment) adaptations. They will also determined sustained effects of the intervention by completing a 9-month follow-up.

DETAILED DESCRIPTION:
The PI will verify age with a drivers license or other form of identification to ensure that the study participants are at least 18 years of age to participate. After obtaining consent, the PI will then administer a pre-exercise screening tool, the Physical Activity Readiness Questionnaire for Everyone, to the participant for them to complete in order to aid in determining study eligibility. If the participant is deemed eligible, 3 other questionnaires will be emailed to participants for completion: Physical Activity Enjoyment Scale, Exercise Self-efficacy Scale, and the International Physical Activity Questionnaire (IPAQ) short form. Given that the participants will be instructed to not change any physical activity habits outside of the study, the IPAQ will be used to control for this pre- and post-intervention and weekly throughout the duration of the intervention. All forms must be completed and submitted to the PI prior to further data collection. Data collection will consist of a (1) blood collection visit, (2) exercise testing and abdominal/visceral fat measurement session, (3) three exercise/movement familiarization sessions (only conducted pre-intervention), (4) three strength, muscular endurance, and muscular power testing sessions before and after the intervention, and 12 weeks of training three times per week as described below. Excluding the consent obtaining meeting, participants will attend 8 sessions prior to beginning the intervention as detailed below. During the intervention, participants will be wearing heart rate monitors in order to monitor their training intensity. The PI will lead all data collection procedures with the assistance of School of Health Science students and Dr. Myung Choi except for the blood collection and analysis which will be supervised by Dr. Kristen Landis-Piwowar. All measures will be assessed pre- and post-intervention. Blind copy emails will be sent to remind the participants about upcoming data collection sessions and to schedule a data collection appointment.

Day 1: Prevention Research Center (blood collection visit)

Following 12-hr fast, assessments include:

* weight, height, waist circumference
* resting heart rate
* blood pressure
* venipuncture (blood sugar and fat)
* blood analysis

Day 2: Prevention Research Center (exercise testing and visceral fat visit)

Assessments include:

* dual-x-ray absorptiometry (DXA) to measure visceral adipose tissue
* bicycle VO2max test with standard warm-up and clinical monitoring to assess aerobic endurance
* Physical Activity Enjoyment Scale and Exercise Self-efficacy Scale (post-intervention)

Days 3-5: Oakland University (OU) Recreation Center (familiarization visits)

Familiarization sessions include:

* teaching movements used in subsequent testing and training
* assessment of musculoskeletal limitations
* intervention leader and assistants will attend sessions as part of training

Days 6-8: OU Recreation Center (performance testing visits)

Assessments include:

* Day 6: one repetition maximum (1 RM) testing for back squat (muscular strength); 70% 1RM back squat for max effort repetitions unbroken (muscular endurance)
* Day 7: 1 RM overhead press (muscular strength)
* Day 8: 1 RM deadlift (muscular strength) and max broad jump (muscular power)
* standardized warm-up prior to cool-down following each session
* at least 48 hours of rest between each session

Pre- and post-intervention health measurements: Prevention Research Center Anthropometrics and vital sign measures such as height (using a stadiometer), weight (using an eye-level beam scale), heart rate and blood pressure (sitting with a sphygmomanometer) will be obtained.

Pre- and post-intervention endurance measurements: Prevention Research Center Aerobic fitness will be directly assessed by a VO2max bicycle test. Each participant will be allowed to warm-up on the bicycle for 5 minutes at a low intensity. The VO2max bicycle test will include 3 minute stages with increasing intensity each stage of 30 - 60 watts. The required cadence will be maintained at 60 revolutions per minute (RPM) for each stage. The test will be terminated at volitional fatigue defined as the participant no longer able to maintain 60 RPMs for 20 seconds after encouragement from the testers. For most people, the test will take approximately 10 minutes.

Pre- and post-intervention strength measurements: OU Recreation Center Prior to strength testing, three familiarization sessions will be conducted whereby participants will be taught and given a chance to practice the movements to be used for testing and training. During these sessions, participants will be assessed for any musculoskeletal limitations such as a lack of hip and ankle mobility that may require movement/exercise modifications to ensure safe technique. Following the familiarization sessions, each participant will complete three further days of testing, with at least 48 hours between testing days. These testing sessions will occur at OU Recreation Center. Each of these test sessions will be preceded by a standardized warmup and instruction regarding the upcoming session. On separate days, muscle strength will be assessed using 1-repetition maximum (1RM) testing for back squat, press, and deadlift using standardized protocols. The back squat will be performed to below parallel (hip crease below the apex of the patella), the press will be initiated with the bar on the clavicles, and the deadlift will performed in the conventional stance. All testing days will be repeated following training.

Pre- and post-intervention muscle endurance and muscle power: OU Recreation Center Muscle endurance will be assessed by repetitive back squats to voluntary exhaustion. The load will be set at 70% of the pre-training

1RM back squat for both pre- and post-training tests. This test will be conducted immediately after the 1 RM testing for back squat. Movement standards will be the same as those for the 1RM test, and the total number of successful repetitions achieved without a rest will be recorded. Muscle power will be assessed using a static broad jump. The best horizontal distance achieved out of 3 trials will be recorded. This test will be conducted immediately after the 1 RM testing for the deadlift.

Pre- and post-intervention biochemistry measurements: Prevention Research Center Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of: total cholesterol, high-density lipoprotein cholesterol, triglycerides, alanine aminotransferase, aspartate aminotransferase, glucose, and low-density lipoprotein cholesterol. This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon). The risks of blood draw may include: infection, delayed healing, bruising and/or inflammation at the site of vein puncture, physical discomfort, mental discomfort, fainting and feeling faint and injury to a nerve or vessel. These risks will be minimized by the use of a trained professional (Dr. Kristen Landis-Piwowar) experienced with performing the blood draws, sterile technique and single use, disposable, materials who will be supervising the blood draw and analysis. Study participants may refuse to participate at any time and withdraw from the study without penalty.

Pre- and post-intervention visceral fat measurement using dual x-ray absorptiometry (DXA) scan: Prevention Research Center For this measurement of visceral fat, each participant will be asked to lie flat on a special table below the DXA scan. A trained technician (Elise Brown, Ryan Tyler, Myung Choi, or Samantha Orr) will position each participant's body under the scan and then perform the scan, which will only take < 5 minutes.

Pre- and post-intervention psychosocial questionnaires The purpose of including these psychosocial assessments in the proposed study is to assess changes in physical activity enjoyment and exercise self-efficacy. High-intensity interval training has been shown to be more enjoyable than continuous training, and this may lead to enhanced self-efficacy. These questionnaires will be emailed to participants for completion: Physical Activity Enjoyment Scale and Exercise Self-efficacy Scale.

Nine months following the intervention, participants will complete all assessments again.

The intervention will be led by students (one leader and at least 2 assistants) who will be trained by the PI, and exercise protocols are as follows:

MM-HIIT Group: This group will train using multimodal exercises for 5 sets of 60 seconds of all out work, followed by 3 minutes of rest (a total of 20 minutes each session). Each session will have the same exercises within each set, but every session will be different than the others for movements utilized. There will be three movements used in each set. The first movement will be a strength movement (such as overhead press, squat, deadlift) for 4-6 repetitions. The second movement follows the first immediately and is a faster body weight or light implement power movement such as lunges, body weight squats, or push ups for 6-8 repetitions. The third movement follows the second immediately and is a very fast, sprint-like movement such as box jumps, ball slams, or jump rope for the remainder of the 60 seconds. The intent of each set is to be completed with as much effort as possible across the full 60 seconds. The intervention leader will record weight used for each exercise and will instruct participants to increase intensity (up to 110% of previous intensity used) at subsequent session once maximum prescribed repetitions have been.

R-HIIT Group: This group will train using a rowing ergometer for 5 sets of 60 seconds of all out work, followed by 3 minutes of rest (a total of 20 minutes each session). Each training session will be the same across the 12 weeks. The intent of each set is to be completed with as much effort as possible across the full 60 seconds.

Control Group: This group will be instructed to continue with any activity they were involved in prior to the study and to not begin any new exercise programs during the course of the study. To incentive participation in this group, the control group will be offered the MM-HIIT intervention the following semester at no cost.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be non-obese (waist circumference ≤ 88 cm) recreationally active females aged 18 - 40 years who do not engage in a regular training program. Recreationally active is defined as periodically participating in physical activity or exercise between 1 - 3 hours a week for at least a month, but not involved in a systematic endurance or weight training activity.

Exclusion Criteria:

* Potential participants will be excluded if they have a history of exercise-limiting cardiovascular, respiratory, metabolic, or musculoskeletal illness/injury or if they are currently taking medication that would alter the physiological responses to exercise. They will also be excluded if they are pregnant or have a history of fainting while giving blood.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Aerobic fitness | 15 minutes
  Aerobic fitness will be directly assessed by a VO2max bicycle test. Each participant will be allowed to warm-up on the bicycle for 5 minutes at a low intensity. The VO2max bicycle test will include 3 minute stages with increasing intensity each stage of 30 - 60 watts. The required cadence will be maintained at 60 RPMs (revolutions per minute) for each stage. The test will be terminated at volitional fatigue defined as the participant no longer able to maintain 60 RPMs for 20 seconds after encouragement from the testers. For most people, the test will take approximately 10 minutes.

SECONDARY OUTCOMES:
Triglycerides | 10 minutes
  Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of triglycerides (mmol/L). This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon).
Physical Activity Enjoyment scale | 5 minutes
  The purpose of including this psychosocial assessment in the proposed study is to assess changes in physical activity enjoyment. Physical Activity Enjoyment Scale

OTHER OUTCOMES:
Muscular Endurance | 5 minutes
  Muscle endurance will be assessed by repetitive back squats to voluntary exhaustion. The load will be set at 70% of the pre-training 1RM back squat for both pre- and post-training tests. The total number of repetitions will be recorded.
Total Cholesterol | 5 minutes
  Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of: total cholesterol (mmol/L), alanine aminotransferase, aspartate aminotransferase, glucose, and low-density lipoprotein cholesterol. This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon).
Visceral Fat | 5 minutes
  For this measurement of visceral fat, each participant will be asked to lie flat on a special table below the DXA scan. A trained technician will position each participant's body under the scan and then perform the scan.
Muscular Strength | 90 minutes
  Each participant will complete three days of testing, with at least 48 hours between testing days. These testing sessions will occur at OU Recreation Center. Each of these test sessions will be preceded by a standardized warmup and instruction regarding the upcoming session. On separate days, muscle strength will be assessed using 1-repetition maximum (1RM) testing for back squat, press, and deadlift using standardized protocols. The back squat will be performed to below parallel (hip crease below the apex of the patella), the press will be initiated with the bar on the clavicles, and the deadlift will performed in the conventional stance. All testing days will be repeated following training.
Muscular Power | 10 minutes
  Muscle power will be assessed using a static broad jump. The best horizontal distance achieved out of 3 trials will be recorded. This test will be conducted immediately after the 1 RM testing for the deadlift.
High-density lipoprotein cholesterol | 10 minutes
  Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of high-density lipoprotein cholesterol (mmol/L). This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon).
Alanine Aminotransferase | 10 minutes
  Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of alanine aminotransferase (U/L). This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon).
Asparate Aminotransferase | 10 minutes
  Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of asparate aminotransferase (U/L). This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon).
Glucose | 10 minutes
  Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of glucose (mmol/L). This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon).
Low-density lipoprotein cholesterol | 10 minutes
  Following a 12-hour fast, participants will complete venipuncture collection procedures. Two invasive needle sticks will be performed during this investigation (one needle stick pre-intervention and another needle stick post-intervention). Four milliliters (mL) of blood will be collected both pre- and post-intervention for measurement of low-density lipoprotein cholesterol (mmol/L). This total amount of blood (8mL) collected during this trial will equate to 1.6 teaspoons of blood (5mL = 1 teaspoon).
Exercise Self-Efficacy Scale | 5 minutes
  The purpose of including this psychosocial assessments in the proposed study is to assess changes in exercise self-efficacy. Exercise Self-efficacy Scale.
Body Mass Index | 1 minutes
  Anthropometrics such as height (cm) using a stadiometer and weight (kg) using an eye-level beam scale will be obtained. Height and weight will then be converted to body mass index (kg/m2)
Weight | 1 minutes
  Anthropometrics such as weight (kg) using an eye-level beam scale will be obtained. Height and weight will then be converted to body mass index (kg/m2)
Height | 1 minutes
  Anthropometrics such as height (cm) using a stadiometer will be obtained. Height and weight will then be converted to body mass index (kg/m2)
Waist Circumference | 5 minutes
  Anthropometrics such as waist circumference (cm) using a Gulick tape will be obtained.
Blood Pressure | 10 minutes
  Vital sign measures such as and blood pressure (mmHg) sitting using a sphygmomanometer will be obtained.
Heart Rate | 2 minutes
  Vital sign measures such as heart rate (bpm) will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Brown, PhD, Principal Investigator — Oakland University
Locations (1):
- Oakland University, Rochester, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rengers TA, Orr SC, Marks CRC, Hew-Butler T, Choi MD, Butcher SJ, Drignei D, Brown EC. Effects of High-Intensity Interval Training Protocols on Liver Enzymes and Wellness in Women. J Sports Med (Hindawi Publ Corp). 2021 Apr 30;2021:5554597. doi: 10.1155/2021/5554597. eCollection 2021. PMID 34007845